CLINICAL TRIAL: NCT03308305
Title: Cracking Coma: Towards EEG and MRI Based Precision Medicine After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: University Medical Center Nijmegen (Other); Donders Centre for Cognitive Neuroimaging (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-1006
Record Dates: First submitted 2017-10-02; First posted 2017-10-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Post-Anoxic Coma; Postanoxic Enchephalopathie
Keywords: Coma; Cardiac arrest; Prognosis; MRI; EEG
MeSH Terms: conditions — Coma; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Of patients who die during ICU stay, families are asked permission for autopsy of the brain. After fixation, multiple fragments of brain tissue will be retained for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: 30-70% of comatose patients admitted to the intensive care unit (ICU) after cardiac arrest never regain consciousness as a result of post anoxic encephalopathy (PAE). Early identification of patients without potential for recovery of brain functioning may prevent inappropriate continuation of medical treatment and improve communication between doctors and patients. However, current diagnostic and prognostic measures can identify only 20-50% of the patients with irreversible brain damage, precluding cerebral recovery and awakening. Also, the pathophysiology of brain damage is largely unclear. New magnetic resonance imaging (MRI) sequences hold potential to substantially improve outcome prediction.

Objectives: 1. To estimate the additional value of early MRI monitoring for the prediction of neurological outcome of comatose patients after cardiac arrest. 2. To gain insight in the pathophysiology of PAE by associating MRI findings with histopathological studies of brain tissue obtained from non-survivors.

Study design: prospective cohort study.

Study population: 100 subsequent comatose patients after cardiac arrest, admitted to the ICU.

Intervention: In addition to standard treatments, patients will undergo MRI of the brain at day 3, 7, and three months after cardiac arrest. A subgroup of patients will be scanned within 24 hours after cardiac arrest, to assess feasibility and to gain more insight in the evolution of brain damage in PAE. Survivors will be followed for one year. Outcome measurements will focus on disabilities, quality of life, and depression. MRI measures will be related to outcome.

Main study parameters/endpoints: The primary outcome measure is neurological outcome, defined as the score on the Cerebral Performance Category (CPC) at six months, dichotomized as good (CPC 1-2 = no or moderate neurological disability) or poor (CPC 3-5 = severe disability, coma, or death). Secondary outcome measures include cognitive functioning, depression, and quality of life at one year, as well as histopathological damage of brain tissue of non-survivors.

DETAILED DESCRIPTION:
Standard procedures:

Patients will be monitored and treated according to guidelines for post out of hospital cardiac arrest treatment as described in local ICU protocols. Patients do not suffer any harm, disadvantage of discomfort while participating in this study.

Standard treatment includes targeted temperature management, hemodynamic monitoring and stabilisation, continuous EEG monitoring, blood sampling through the jugular bulb catheter, Near Infrared Spectroscopy (NIRS), and transcranial doppler (TCD) measurements. The patient's status is repeatedly assessed and treatment is based on the clinical findings.

Additional procedures:

1. MRI A total of 3 MRI scans is planned for each patient: at day 3 ± 1, and day 7 ± 2 after cardiac arrest, and 3 months ± 2 weeks after cardiac arrest. The imaging protocol will consist of structural MRI (including FLAIR and ADC maps) to detect ischemic damage, a 3D T1 for structural analysis and SWI sequences to detect micro bleeds), structural connectivity measurement by DTI, and functional connectivity measurement by resting state BOLD functional MRI. Estimated time to prepare the patient and transport to and from the MRI scanner will be approximately 30 minutes, the scan itself will take approximately 30 minutes, as well. No intravenous contrast agent is used.

   1.1 Acute phase MRI To estimate the feasibility of MRI scanning in the acute phase and to gain more insight in the dynamics of PAE, a subgroup of patients will be scanned within 24 hours after cardiac arrest. Patients will be included in this subgroup dependent on availability of the MRI facility, the clinical stability of the patients and after the patients legal representatives signed informed consent.

   1.2 Transport to the radiology department

   The transport to and from the radiology department will be performed as described in the local protocols on patient transportation. Transport to and from other departments is a frequent procedure in ICU patients. During transport, the patient will be accompanied by a physician and ICU nurse. The MRI scans for this project will be handled as 'elective', which indicates that only patients with a stable hemodynamic and respiratory status will be transported to and undergo the MRI. For this, a patient has to meet all the following criteria:

   A. Hemodynamic stable condition, defined as:
   * mean arterial pressure > 60 mmHg
   * no or low inotropes or vasopressors (dosage norepinephrine < 0,3 ug/kg/min and/or dobutamine < 10 ug/kg/min or equivalent), dosage adjustments less than 0.1 ug/kg/min in the last hour before MRI

   B. Stable cardiac rhythm, defined as:
   * sinus rhythm 50 - 120 beats per minute
   * atrial fibrillation or flutter with ventricle response 60 - 120 per minute

   C. Pulmonary stable condition, defined as:
   * Arterial oxygen saturation > 95%
   * maximum fraction inspired oxygen < 60% with maximum level of positive end expiratory pressure of 10 cm H2O
   * peak inspiratory pressure < 30 cmH2O or <5 l/min oxygen trough nasal cannula (for patients not on mechanical ventilation)

   Mechanical ventilation during transport and scanning will be provided by an MRI compatible ventilator.

   Extensive monitoring of vital functions will not be interrupted during transport or MRI scanning, by using a mobile trolley with MRI compatible monitoring and ventilation equipment. At all times, a physician and trained ICU nurse will accompany the patient. The medical team accompanying the patient can change treatment during transport and scanning to pursue optimal hemodynamics, pulmonary state, and/or comfort.

   1.3 Clinical evaluation of MRI scans All structural MRI scans will be assessed by a radiologist and results are added to a patient's medical file. Patients and their families will be informed. However, MRI findings will not be taken into account for decisions on withdrawal of treatment. BOLD fMRI and DTI data will be analysed later.
2. Outcome At 3 and 6 months, CPC score will be assessed by a telephone interview by a trained investigator. Additionally, at twelve months, for assessment of cognitive outcome, depression, quality of life, and care giver strain, the patient will be invited to the hospital or visited at his / her place of residence. If a patient dies during the follow-up, the cause of death will be requested from the general practitioner or medical specialist.
3. Post mortem analysis From all patients that die in the hospital after PAE, permission to perform autopsy is sought for. Permission will be asked from the legal representative in the context of current care, after the patient has died. According to current care, brains will be removed and samples fixated within 24 hours at the local pathology departments. On samples from 8 brain areas (sensory- and motor cortex, thalamus, basal ganglia, upper brain stem) evaluation of the agonal state is performed on hematoxylin-eosin staining. Additionally, predefined sections, including all cortical layers and white matter, will be formalin fixed for further analyses.

ELIGIBILITY:
Inclusion Criteria:

* Comatose, defined as Glasgow Coma Score ≤ 8
* Age ≥ 18 years
* Cardiac arrest with a presumed cardiac cause of the arrest or caused by pulmonary embolism
* Admission to ICU

Exclusion Criteria:

* Pregnancy
* Life expectancy < 24 hours
* Absence of written informed consent (by a legal representative)
* Pre-existing dependency in daily living, defined as CPC score 3 or 4
* Any known progressive brain illness, such as a brain tumor or neurodegenerative disease.
* Known contra-indication for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of one hundred adult, comatose patients, successfully resuscitated from cardiac arrest. Generally, these patients are predominantly male and approximately 60-65 years of age. The patients are by definition at least temporarily incapacitated.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Functional outcome | 6 months after cardiac arrest
  Functional outcome as defined on the Cerebral Performance Category , dichotomized as good (CPC 1-2 = no or moderate neurological disability) or poor (CPC 3-5 = severe disability, coma, or death)

SECONDARY OUTCOMES:
cognitive functioning as defined by professional Neuropsychological examination | 12 months after cardiac arrest
  By using a standardized Neuropsychological examination, the cognitive state of a patient will be assessed one year after the cardiac arrest. The examination will focus on memory, language, executive functioning, speed of information processing, concentration and attention and visuoconstruction.
Presence of depression | 12 months after cardiac arrest
  Presence of depression is scored using a Dutch translation of the HADS questionnaire.
histopathological damage of brain tissue of non-survivors | Autopsy will take place at the first workday after the patient died at the ICU after cardiac arrest. After 2 weeks, the brain will be cut and paraffine coupes will be made. Analyses of the coupes will take place in batches.
  After fixation, histopathological staining will be performed on gray matter and white matter structures of the brain. Different stainings will be used to asses morphological damage, synaptic damage and membrane damage.
Early functional outcome | At discharge from the ICU and 3 months after cardiac arrest.
  Functional outcome as defined on the Cerebral Performance Category, scored at discharge from the ICU and 3 months after cardiac arrest
Participation in society score | 12 months after cardiac arrest
  The USER-Participate questionnaire will be used to evaluate a subjects participation in society.
EQ-5D-5L quality of life | 12 months after cardiac arrest
  Quality of life will be scored by the EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: J Hofmeijer, PhD, Principal Investigator — Rijnstate Hospital
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Radboud University Medical Centre, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Verhulst MMLH, Keijzer HM, van Gils PCW, van Heugten CM, Meijer FJA, Tonino BAR, Bonnes JL, Delnoij TSR, Hofmeijer J, Helmich RC. Functional connectivity in resting-state networks relates to short-term global cognitive functioning in cardiac arrest survivors. Hum Brain Mapp. 2024 Oct 15;45(15):e26769. doi: 10.1002/hbm.26769. PMID 39449030
- [Result] Keijzer HM, Duering M, Pasternak O, Meijer FJA, Verhulst MMLH, Tonino BAR, Blans MJ, Hoedemaekers CWE, Klijn CJM, Hofmeijer J. Free water corrected diffusion tensor imaging discriminates between good and poor outcomes of comatose patients after cardiac arrest. Eur Radiol. 2023 Mar;33(3):2139-2148. doi: 10.1007/s00330-022-09245-w. Epub 2022 Nov 24. PMID 36418623
- [Result] Keijzer HM, Lange PAM, Meijer FJA, Tonino BAR, Blans MJ, Klijn CJM, Hoedemaekers CWE, Hofmeijer J, Helmich RC. MRI markers of brain network integrity relate to neurological outcome in postanoxic coma. Neuroimage Clin. 2022;36:103171. doi: 10.1016/j.nicl.2022.103171. Epub 2022 Aug 26. PMID 36058165
- [Result] Keijzer HM, Verhulst MMLH, Meijer FJA, Tonino BAR, Bosch FH, Klijn CJM, Hoedemaekers CWE, Hofmeijer J. Prognosis After Cardiac Arrest: The Additional Value of DWI and FLAIR to EEG. Neurocrit Care. 2022 Aug;37(1):302-313. doi: 10.1007/s12028-022-01498-z. Epub 2022 Apr 25. PMID 35469391